CLINICAL TRIAL: NCT06960941
Title: Evaluation of the Effect of Dietary Supplementation With Probiotics and Prebiotics on Inflammatory Processes, Motor and Cognitive Performance in Patients With Gastrointestinal Disorders.
Brief Title: Evaluation of Dietary Supplementation in Patients With Gastrointestinal Disorders.
Acronym: TrioB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7272
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome; Metabolic Syndrome
Keywords: Inflammation; Irritable Bowel Syndrome; Metabolic Syndrome; Nutrition
MeSH Terms: conditions — Irritable Bowel Syndrome; Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G-TrioB (Experimental): G-TrioB patients, without making any changes to his or her current medication routine, if any, will take 1 sachet of TrioBiotiotix360® daily for 3 months (12 weeks) and will receive a pamphlet with a series of postural hygiene exercises to be performed at home (at least 30 minutes a day, 5 days a week).
  Interventions: Dietary Supplement: TrioBiotix360®; Other: Booklet with a series of postural hygiene exercises
- G-CON (Active Comparator): G-CON patients will only receive a booklet with a series of postural hygiene exercises to be performed at home (at least 30 minutes a day, 5 days a week) for a period of 3 months.
  Interventions: Other: Booklet with a series of postural hygiene exercises

INTERVENTIONS:
Dietary Supplement: TrioBiotix360® — Dietary supplement combining prebiotics and probiotics to promote the balance of intestinal bacterial microflora.
  Arms: G-TrioB
Other: Booklet with a series of postural hygiene exercises — The booklet will contain a series of postural hygiene exercises to be performed at home

SUMMARY:
The term "inflammaging" describes the aging process characterized by a chronic low-grade inflammatory state. With advancing age, this condition is often associated with cardiovascular disease, diabetes, and neurodegenerative diseases. Often, the inflammaging state is characterized by environmental factors, such as pollution, diet, and physical inactivity, as well as the accumulation of free radicals and alteration of the gut microbiota. Inflammaging also appears to be linked to irritable bowel syndrome (IBS), a functional gastrointestinal disorder characterized by chronic abdominal pain and altered bowel habits, and is related to low-grade mucosal inflammation, which may contribute to visceral hypersensitivity and symptom severity.In addition, cytokine activity and alterations in intestinal immune cells would appear to participate significantly in the pathogenesis of IBS. Additionally, there is an independent correlation between IBS and a higher prevalence of metabolic syndrome. Given the multifactorial nature of IBS, no effective treatment has been identified to date. However, considering the central role that alteration of the gut microbiota plays in IBS, the use of prebiotics and probiotics may represent an alternative therapy, as well as help in managing the inflammatory state. Probiotics are live organisms present in the intestinal tract that have the ability to resist the action of digestive enzymes.

DETAILED DESCRIPTION:
Probiotics such as Lactobacillus and Bifidobacterium can interact with immune cells, promoting the synthesis of anti-inflammatory cytokines such as IL-10. Studies have shown that they can significantly reduce inflammatory markers such as TNF-α and C-reactive protein (CRP) in conditions such as nonalcoholic hepatic steatosis.

Prebiotics, on the other hand, are substances that are not digestible by the body and are intended to assist the function of probiotics: prebiotics such as β-frucans and galacto-oligosaccharides selectively stimulate beneficial gut bacteria, which can attenuate inflammation in inflammatory bowel disease models. In addition, the production of short-chain fatty acids from prebiotic fermentation is linked to the reduction of systemic inflammation, as shown by decreased CRP levels in subjects consuming different prebiotic mixtures.

The combined use of probiotics and prebiotics, in addition to modulating inflammation, could also influence motor and cognitive function. Recent studies have demonstrated the beneficial effects of probiotics and prebiotics on coordination and motor function in various models, including Parkinson's disease.

Patients referred to the UOS Post-Acute Rehabilitation, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, who meet the inclusion criteria will be recruited. Patients will be randomly divided into two groups as specified below. One group (G-TrioB), without making any changes to the current therapeutic routine, will take 1 sachet of TrioBiotix360® daily for 3 months (12 weeks) and will receive a pamphlet with a series of postural hygiene exercises to be performed at home (at least 30 minutes per day, 5 days per week); the other group (G-CON) will receive only a pamphlet with a series of postural hygiene exercises to be performed at home (at least 30 minutes per day, 5 days per week) for a period of 3 months.

In addition, studies have shown the effect of probiotics on cognitive function, particularly in individuals with mild cognitive impairment and Alzheimer's disease; prebiotics, by enhancing the efficacy of probiotics, may promote a favorable environment for the gut microbiota, which is critical for cognitive health.

Triobiotix360® is a dietary supplement that combines prebiotics and probiotics to support the balance of intestinal bacterial microflora. The prebiotic component is characterized by the presence of Bioecolicans® gluco-oligosaccharide fiber, while the probiotic component is characterized by the presence of Bifidobacterium animalis ssp. Lactis BLC1 (DSM 17741), Lactobacillus acidophilus LA3 (DSM 17742), Lactobacillus rhamnosus IMC 501 (DSM 16104), Lactobacillus paracasei IMC 502 (DSM 16105) and Streptococcusther-mophilus SP4 (DSM 19385). This effect is enhanced by the presence of hyaluronic acid and a mineralized extract of Lithothamnion, a source of calcium, which contributes to the normal functioning of digestive enzymes. Innovative T_win packaging technology preserves the viability of the mixture of 5 different starter culture bacterial strains, selected and blended to maximize product functionality.

ELIGIBILITY:
Inclusion Criteria:

* At least two criteria required for the diagnosis of IBS, according to Rome IV criteria (Lacy et al., 2021), namely:

  * presence of recurrent abdominal pain on an average of at least 1 day per week in the past 3 months, associated with two (or more) of the following criteria:
  * Related to defecation;
  * Associated with a change in stool frequency;
  * Associated with a change in stool shape/appearance.
* At least two criteria required for the diagnosis of metabolic syndrome, namely:

  * impaired blood glucose/insulin resistance;
  * Central obesity, waist/hip ratio > 0.9 in males; > 0.85 in females; and/or Body Mass Index (BMI) >30;
  * blood pressure ≥ 160/90 or taking antihypertensive drugs;
  * HDL cholesterol < 35 mg/dl in males; < 39 mg/dl in females;
  * triglycerides ≥ 150 mg/dl;
  * microalbuminuria > 20μg/min or albumin/creatinine ratio > 20mg/g (presence of trace amounts of albumin in urine.

Exclusion Criteria:

* Hypersensitivity to one or more ingredients;
* Diagnosis of metabolic syndrome;
* Prior history of stroke and/or myocardial infarction;
* Presence of altered mood;
* Presence of kidney or intestinal disease, pancreatitis, diabetes, or any other endocrine disorder;
* Presence of demyelinating and dysmyelinating diseases;
* Inability to provide informed consent.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
CRP | Change from Baseline PCR at 3 months and at 6 months
  C-reactive protein (CRP) is an index of inflammation; as such, its blood concentrations increase in the presence of inflammatory processes of various types.
  CPR cutoffs are 0-0.5 mg/dL, absence of inflammatory processes; 0.5-1.0 mg/dL, non-acute inflammatory state; 1.0-10 mg/dL: mild or moderate acute inflammation; > 10 mg/dL, extensive inflammation

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 3 months and at 6 months
  SPPB is an objective measurement instrument of balance, lower lowerextremity strength, and functional capacity in older adults (>65 years of age). Three domains, which include balance, usual or self-selected gait speed, and lower limb strength, are assessed by a three-stage balance test (feet side-by-side, semitandem, and tandem positions), a 3-m or 4-m gait speed test (time spent to walk the course), and a repetitive chair stand test (five times chair sit-to-stand test), respectively. A 0- to 12-point scale is used to score the sum of the three assessments, with point values corresponding with greater levels of function and lower disability, whereas lower point values correspondwith lower levels of physical function and higher disability, respectively
Timed 25 Foot Walk (T25FW) | Change from Baseline T25FW at 3 months and at 6 months
  The T25-FW is a quantitative test of leg mobility and function based on a timed 25-foot walk. The patient is directed to one end of a path and instructed to walk as quickly but safely as possible. The task is immediately repeated by asking the patient to return by walking the same distance. Patients may use assistive devices while performing this task.
Timed Up&Go Test (TUG) | Change from Baseline TUG at 3 months and at 6 months
  TUG measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down.
  The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 5is severely abnormal) according to the observer's perception of the patient's risk of falling.
  The timed part of the test records the mean time (in seconds) from frominitial getting up to re-seating. Patients are compared with the mean time of adults in their age group: 60 to 69, 70 to 79, and 80 to 99 years of age.
Trail Making Test (TMT) | Change from Baseline TMT at 3 months and at 6 months
  The TMT measures flexibility of thinking on a visual-motor sequencing task. It consists of two parts, A and B, where 25 circles are distributed over a sheet of paper. In Part A, the circles are numbered 1-25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1-13) and letters (A-L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
  Trail A: Average 29 seconds, Deficient > 78 seconds, Rule of most in 90 seconds Trail B: Average 75 seconds, Deficient > seconds, Rule of Thumb Most in 3 minutes
Symbol Digit Modalities Test (SDMT) | Change from Baseline SDMT at 3 months and at 6 months
  The SDMT is a neuropsychological test used to assess cognitive processing speed, attention, and visual-motor coordination. The test involves matching symbols to corresponding numbers based on a key, and participants must quickly and accurately pair the symbols with the correct numbers within a set time limit.
  The test evaluates attention, working memory, and mental flexibility. A higher score indicates better cognitive processing speed and accuracy.
Stroop Colour Word Test (SCWT) | Change from Baseline SCWT at 3 months and at 6 months
  ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. The subject is asked to read the words in the first task and to name colors in the second and third tasks. It is necessary to mark not only any mistakes made but also the time spent on each task. The cut-off for the error interference effect is 4.24, while the cut-off for the time interference effect is 36.92.
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline HADS at 3 months and at 6 months
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale, the score is the sum of the respective seven items (ranging from 0 to 21).
  The two sub-scales, anxiety and depression, have been found to be beindependent measures. In its current form, the HADS is now divided into four stages:
  Scores of 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 3 months and at 6 months
  The MFIS is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items, while the abbreviated version has 5 items.
  The MFIS is a structured, self-report questionnaire that the patient can cangenerally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.
EuroQoL- 5D (EQ-5D) | Change from Baseline EQ-5D at 3 months and at 6 months
  EQ-5D is an instrument that evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to the ED-5D permit finding 243 unique health states or can be converted into EQ-5D index and utility scores anchored at 0 for death and 1 for perfect health.
Irritable Bowel Syndrome-Quality of Life (IBS-QOL) | Change from Baseline IBS-QOL at 3 months and at 6 months
  The IBS-QOL is a self-assessment tool for quality of life. The IBS-QOL consists of 34 items, each with a five-point response scale: from 1 (not at all) to 5 (very much).
  Individual responses to the 34 questions are summed and averaged to obtain a total score, which is then transformed into a scale of 0 to 100 for ease of interpretation, where higher scores indicate better quality of life.
Silver Index (SI) | Change from Baseline SI at 3 months and at 6 months
  The SI is an objective test to identify the risk of falling, which is carried out using the Hunova robotic platform. It consists of seven domains:
  (i) static balance (ii) dynamic balance (iii) reactive balance (iv) sensory sensoryintegration (v) stability limits (vi) sitting-to-standing position (vii) gait speed.
  At the end of the evaluation, you get a percentage that indicates risk of falling
Bioimpedance analysis (BIA) | Change from Baseline BIA at 3 months and at 6 months
  BIA measures the opposition of body tissues to alternating current, that is, the impedance of the whole body. The two raw parameters derived from this analysis are resistance (Rz) and reactance (Xc). Rz is inversely related to water content in biological tissues, while Xc depends on the capacitance properties of the cell membrane, providing information on cellular health, integrity, and density From Rz and Xc, the phase angle (PhA), which is related to cellular health and muscle quality, can be calculated directly.
  Lower PhA values have typically been observed in subjects with severe pathological conditions and have been correlated with worse outcomes; in contrast, higher PhA values are indicative of better overall health, strength, and muscle function.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy